CLINICAL TRIAL: NCT04650373
Title: Long-term Durability of Weight Loss After Bariatric Surgery; A Retrospective Study
Brief Title: Durability of Weight Loss After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdulkarim Hasan, Pathologist and Laboratory Director, Al-Azhar University
Other Study IDs: AUH20-011
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Obesity
Keywords: Bariateric surgery; Durability
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical management: Underwent bariatric surgery
  Interventions: Procedure: Bariateric surgery
- Non-surgical management: Patients treated medically

INTERVENTIONS:
Procedure: Bariateric surgery — Adult patients underwent RYGB surgical treatment during the period from 2014 to 2019
  Groups: Surgical management

SUMMARY:
The present study is a retrospective cohort study. Patients older than 18 years of age and underwent Roux-en-Y gastric bypass (RYGB) surgical treatment during the period from 2014 to 2019 and paired severely overweight controls who had no longer gone through bariatric surgery. Patients having BMI (Body Mass Index) much lower than 35 (calculated as the weight (kilograms) / length2 (meters)), a base line diagnosis taken into consideration a medical exclusion for surgical treatment died in one year of surgical operation and missed statistics at scientific information had been excluded from the study. The primary final results of the study was the weight-change percentage at follow-up in comparison with baseline one and the clinical events after surgery.

DETAILED DESCRIPTION:
This is a retrospective cohort study. The sample size of our study includes one hundred case older than 18 years of age and underwent RYGB surgical treatment during the period from 2014 to 2019 and paired severely overweight controls who had no longer gone through bariatric surgery. Patients having BMI (Body Mass Index) much lower than 35 (calculated as the weight (kilograms) / length2 (meters)), a base line diagnosis taken into consideration a medical exclusion for surgical treatment, died in one year of surgical operation and missed statistics at scientific information had been excluded from the study. Data was collected taking in to account each patient history (age, sex, length, weight, BMI, occupation, marital status, and comorbidities) and weight record in every visit from measurements statistics. Outcomes: The primary final results of the study was the weight-change percentage at follow-up in comparison with baseline one. The secondary effects including the clinical events after surgery, micronutrient levels, incidence of diabetes, hypertension, and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients equal or over 18 years old
* BMI more than 40
* Complete follow up

Exclusion Criteria:

* No complete follow up
* Age less than 18 or more than 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Al-Azhar University hospital for overweight or obesity problems
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01-17 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
weight-change percentage at follow-up | 1 year
  Weight loss or gain in kilogram after surgery is evaluated.
Clinical Events, Diabetes Miletus | 1 year
  The secondary effects of the clinical events after surgery including incidence of diabetes disease (DM) is measured using the blood glucose level. Fasting blood glucose level more than 7.1 mmol/L is considered posutive for DM
Clinical Events, Hypertension | 1 year
  Arterial blood pressure is followed up regularly, three consequences increase of the blood pressure more than 140 mm Hg systolic and 90 mm Hg diastolic, is positive for hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Baheeg, Study Chair — Al-Azhar University
Locations (1):
- Abdulkarim Hasan, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided